CLINICAL TRIAL: NCT00912899
Title: A Phase I Open Label Study of Noscapine HCl (CB3304 ) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Noscapine HCl (CB3304 ) in Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated early due to lack of clinical response.
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COU-NOS-001
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Refractory Multiple Myeloma
Keywords: Refractory Multiple Myeloma; CB3304; Noscapine HCl; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Noscapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One (Experimental): Noscapine HCl
  Interventions: Drug: Noscapine HCl

INTERVENTIONS:
Drug: Noscapine HCl — Escalating doses given twice per day
  Other Names: Noscapine HCl (CB3304)

SUMMARY:
This is a phase 1 study to evaluate the safety and determine maximum tolerated dose, safety & tolerability of noscapine HCl in patients with advanced multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Advanced Multiple Myeloma.
* Progression after ≥ 2 lines of prior therapy, including at least one steroid, one immunomodulatory agent (iMID), one alkylator, and bortezomib (VELCADE®).
* ECOG performance status of either 0 or 1.

Exclusion Criteria:

* Prior chemotherapy with antimicrotubule agents
* Metastasis involving the brain or spinal cord
* Clinically significant lung or heart disease
* Abnormal electrocardiogram

Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose | During the first 28 day treatment cycle

SECONDARY OUTCOMES:
To determine the safety and tolerability in the study population | End of the study treatment
To evaluate the pharmacokinetics of study drug | End of the study treatment
To assess anti-tumor effects as classified by International Uniform Response Criteria for Multiple Myeloma | End of the study treatment

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Columbia Presbyterian Hospital, New York, New York

REFERENCES:
- See also: NATIONAL CANCER INSTITUTE — http://www.cancer.gov/
- See also: MEDLINE PLUS — http://www.nlm.nih.gov/medlineplus/medlineplus.html
- See also: MULTIPLE MYELOMA — http://www.nlm.nih.gov/medlineplus/multiplemyeloma.html